CLINICAL TRIAL: NCT04369209
Title: A Registered Observational Cohort Study of Facioscapulohumeral Muscular Dystrophy Type 1
Brief Title: A Registered Cohort Study on FSHD1
Status: Recruiting | Type: Observational
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., Professor, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Other Study IDs: MRCTA,ECFAH of FMU [2020]026
Record Dates: First submitted 2020-04-26; First posted 2020-04-30 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Facioscapulohumeral Muscular Dystrophy Type 1 (FSHD1)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The data to be collected is intended to help healthcare providers make important medical and financial decisions concerning FSHD1, through an enhanced understanding of the prevalence, progression and natural history of FSHD1.

DETAILED DESCRIPTION:
The China FSHD1 patient registry is a nationwide, population-based, non-interventional, observational cohort clinical study of all age groups of genetically-confirmed FSHD1 patients from families (with at least 1 affected member), collecting data retrospectively at study entry and prospectively during follow up. The data to be collected is intended to help healthcare providers make important medical and financial decisions concerning FSHD1, through an enhanced understanding of the prevalence, progression and natural history of FSHD1.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of all ages at baseline
* Subjects, with or without symptoms, with FSHD1 genetic confirmation through PFGE-based Southern blotting
* Unrelated healthy controls

Exclusion Criteria:

* Decline to participate
* Other neuromuscular disease (such as Limb-girdle muscular dystrophy or Myotonic dystrophy)
* Serious systemic illness (such as heart, liver, kidney disease or major mental illness)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All genetically-confirmed FSHD1 patients from families (with at least 1 affected member) in China, irrespective of age. These FSHD1 patients presented at least one contracted D4Z4 repeats with 4qA-specific FSHD1-permissive haplotype, the diagnosis of which was performed at Fujian Neuromedical Center (FNMC), the clinical genetic test hospital for FSHD1 in China to employ PFGE-based Southern blotting.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-01 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
PFGE-based Southern blotting | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  Genetic test of PFGE-based Southern blotting were performed for these clinical suspected FSHD1 patients on the basis of the family as a whole. Eligible participants were genetically confirmed patients who presented a contraction to 1-10 D4Z4 repeats with a 4qA-specific FSHD1-permissive haplotype.
The FSHD Clinical Score | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  The FSHD Clinical Score was used to define numerically the clinical severity of facioscapulohumeral muscular dystrophy (FSHD), which was divided into six independent sections that assess the strength and the functionality of (I) facial muscles (scored from 0 to 2); (II) scapular girdle muscles (scored from 0 to 3); (III) upper limb muscles (scored from 0 to 2); (IV) distal leg muscles (scored from 0 to 2); (V) pelvic girdle muscles (scored from 0 to 5); and (VI) abdominal muscles (scored from 0 to 1).

SECONDARY OUTCOMES:
The modified Medical Research Council (MRC) scale | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  The modified Medical Research Council (MRC) scale was used to assess numerically the muscle strength of FSHD participants. Firstly, muscles were tested bilaterally (when applicable) in standardized positions with manual muscle testing (MMT) scores. Then, MMT scores were converted to calculable data of the modified MRC scale.
The Comprehensive Clinical Evaluation Form (CCEF) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 years
  The 2016 Comprehensive Clinical Evaluation Form (CCEF) for FSHD was used to classify phenotypes: category A , typical penetrant patients with both facial and upper limb muscle weakness (subcategories A1: severe facial weakness; A2, moderate facial weakness; A3: only upper or lower facial weakness); category B, atypical penetrant patients (subcategories B1, muscle weakness limited to scapular girdle; B2, muscle weakness limited to facial); category C, asymtomatic (subcategories C1) or nonpennetrant (subcategories C2) patients; and category D, subjects with myopathic phenotype not consistent with FSHD canonical phenotype.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT04369209/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT04369209/ICF_001.pdf